CLINICAL TRIAL: NCT03643055
Title: Diagnostic Value of 18F-Fluorocholine PET/CT for the Detection of Medullary Thyroid Cancer
Brief Title: 18F-Fluorocholine PET/CT in Medullary Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Institute of Oncology Ljubljana (Other)
Responsible Party: Principal Investigator, Luka Lezaic MD PhD, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: 92/08/14
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Medullary Thyroid Cancer
Keywords: medullary thyroid cancer; imaging; hybrid-imaging; 18F-choline; 18F-fluorocholine; PET; PET/CT
MeSH Terms: conditions — Carcinoma, Medullary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MTC 18F-fluorocholine PET/CT: Patients with medullary thyroid cancer imaged using 18F-fluorocholine PET/CT.
  Interventions: Diagnostic Test: 18F-fluorocholine PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-fluorocholine PET/CT — 18F-fluorocholine PET/CT imaging of the neck, mediastinum and whole body.

SUMMARY:
To assess the diagnostic accuracy of 18F-Fluorocholine PET/CT for the detection of medullary thyroid cancer in patients with primary and recurrent disease.

DETAILED DESCRIPTION:
Medullary thyroid cancer (MTC) is a relatively rare type of cancer that represents up to 10% of all primary thyroid cancers. It is a neuroendocrine tumour derived from parafollicular C-cells of the thyroid. It occurs either sporadically or in a hereditary form as a component of the type 2 multiple endocrine neoplasia (MEN) syndromes, MEN2A and MEN2B, and the related syndrome, familial MTC (FMTC).

Currently, the diagnosis of MTC is suspected based on the results of fine-needle aspiration (FNA) cytology, immunohistochemical analysis and elevated laboratory values of tumour markers calcitonin (Ctn) and carcinoembryonic antigen (CEA). According to the 2015 ATA guidelines, the preoperative imaging workup in all patients should include ultrasound examination of the neck; in selected patients, contrast-enhanced CT of the neck and chest, three-phase contrast-enhanced multi-detector liver CT, or contrast-enhanced MRI of the liver, and axial MRI and bone scintigraphy is also recommended. The curative therapy of choice is surgical removal of the tumour and/or metastases.

Nodal metastases are detected in 35-50% and distal metastases in about 15% of patients with primary MTC. Even with currently recommended diagnostic imaging techniques, about 50% of patients have persistent/recurrent disease after surgical treatment. This implies that currently available diagnostic imaging studies are suboptimal for accurate disease staging. New hybrid molecular imaging techniques based on SPECT/CT and especially PET/CT could improve disease detection by visualising pathophysiological processes in vivo. The most studied PET radiopharmaceutical for MTC imaging to date has been 18F-FDOPA, with recent studies focusing also on somatostatin receptor imaging using 68Ga-DOTATATE/TOC/NOC radiotracers.

18F-fluorocholine is a structural analogue of choline. It accumulates in cells with active membrane synthesis and overexpressed intracellular signal transduction, processes that are overactive in benign and malignant neoplasms. 18F-fluorocholine is currently primarily used for prostate cancer imaging. In contrast to radiotracers such as18F-fluorodeoxyglucose (18F-FDG), it is also taken up by well-differentiated neoplasms in which 18F-FDG uptake is unreliable. Similarly to 18F-FDG, 18F-fluorocholine is also known to accumulate in inflamed and infected tissue. However, this limitation could be overcome by performing multi-time-point imaging and using basic kinetic analysis. The working hypothesis is that 18F-fluorocholine might be efficiently taken up by primary MTC tumour as well as loco-regional and distant metastases.

The aim of the trial is to investigate the diagnostic accuracy of 18F-fluorocholine PET/CT in comparison to existing imaging modalities (US, CT and MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with medullary thyroid cancer (sporadic or hereditary form).
* Patients with newly diagnosed MTC for primary staging (based on fine needle aspiration cytology results).
* Patients with suspicion of MTC recurrence for re-staging (based on biochemical, conventional imaging or clinical examination).
* Patients with metastatic MTC on systemic therapy for disease activity assessment.

Exclusion Criteria:

* Pregnancy.
* Patient with any PET/CT-scan exam contraindication (eg. severe claustrophobia).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with medullary thyroid cancer treated at the Institute of Oncology Ljubljana.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-09-03 (Actual); Primary Completion 2021-03-03 (Estimated); Study Completion 2024-09-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy in primary medullary thyroid cancer | 1 month
  Ability to detect primary medullary thyroid cancer (primary, nodal and metastatic lesions) in correlation with histopathological and/or conventional imaging data.
Sensitivity, specificity, positive predictive value, negative predictive value and diagnostic accuracy in recurrent medullary thyroid cancer | 3 months
  Ability to detect recurrent medullary thyroid cancer (nodal and distant metastatic lesions) in correlation with histopathological and/or conventional imaging data.

SECONDARY OUTCOMES:
Survival analysis based on the initial PET/CT examination | 5 years
  Survival analysis of the time to disease progression or disease recurrence after the initial PET/CT examination.
Biochemical/clinical outcome - Ctn levels | 5 years
  Normalization/stable elevation/increasing levels of serum Ctn.
Biochemical/clinical outcome - CEA levels | 5 years
  Normalization/stable elevation/increasing levels of serum CEA.
Correlation between tumour metabolic activity and biochemical and histological markers | 1 month
  Correlation of tumour metabolic activity with biochemical serum marker levels (Ctn, CEA) and tumour metabolic activity and histological quantitative indexes (eg Ki-67).
Modification rate of patient's surgical and medical care after 18F-fluorocholine PET/CT | 5 years
  Rate of patients whose management was modified based on the PET/CT imaging findings.
Basic kinetic analysis of metabolic activity in the primary tumour, nodal and distant metastases. | 3 months
  Ability to differentiate benign and malignant lesions using multiple-time-point imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Department for nuclear medicine, University medical centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided